CLINICAL TRIAL: NCT06142422
Title: Intermittent Theta Burst Stimulation of the Precuneus for the Treatment of Resistant Schizophrenia
Brief Title: Intermittent Theta Burst Stimulation of the Precuneus
Acronym: Stim-TISiTBS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Collaborators: Euraxi Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-A01006-39
Record Dates: First submitted 2023-11-16; First posted 2023-11-21 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: interventional, prospective, randomized, double-blind, multicenter study
Who Masked: Participant, Investigator
Masking Description: Remote coil change while keeping the patient and investigator blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group with intermittent Theta Burst Stimulation (Experimental): The procedure under study is the use of a stimulation device to perform intermittent Theta Burst Stimulation treatment on the precuneus to treat resistant schizophrenia. Targeting requires a neuronavigation device.
  Interventions: Procedure: stimulation device
- control group with placebo stimulation (Placebo Comparator): In the control group, stimulation is simulated using a "Sham" or placebo coil. The stimulation device is the same as for the experimental group, only the coil differs.
  Interventions: Procedure: stimulation device

INTERVENTIONS:
Procedure: stimulation device — The procedure under study is the use of a stimulation device to perform treatment on the precuneus to treat resistant schizophrenia in patients exposed to childhood trauma.
  The target is the left precuneus, which is defined by neuronavigation.

SUMMARY:
The purpose of the study is to compare the effectiveness of stimulation of the left precuneus by intermittent Theta Burst Stimulation to placebo stimulation on the severity of schizophrenia symptoms.

DETAILED DESCRIPTION:
This is an interventional, prospective, randomized, double-blind, multicenter study, comparing iTBS treatment (experimental group) of the precuneus to placebo stimulation (control group) of patients suffering from resistant schizophrenia and having been exposed to childhood trauma.

The study population will be patients aged 18 to 40 years old exposed to childhood trauma, presenting with schizophrenia resistant to antipsychotic treatments.

This study will be implemented in 4 investigative centers. Each patient will participate for a period of 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed patient aged 18 to 40 years inclusive;
* Patient presenting schizophrenia as defined in the Diagnostic and Statistical Manual-5;
* Patient under antipsychotic treatment in accordance with the recommendations of the High Authority of Health, at a stable dosage and without modification of psychotherapeutic treatment for at least 4 weeks;
* Patient on mono or dual antipsychotic therapy.
* Patient presenting residual symptoms, i.e. absence of remission defined by the criteria of the "Remission criteria of the Schizophrenia Working Group Consensus";
* Patient having been exposed to at least one type of trauma in childhood and having a score higher than the threshold values of the childhood trauma questionnaire: emotional neglect, physical abuse, emotional abuse, physical neglect, sexual abuse;
* Patient having signed an informed consent form to participate in the study.

Exclusion Criteria:

* Patient with a contraindication to magnetic resonance imaging or intermittent Theta Burst Stimulation (presence of a metallic body, pacemaker, implantable defibrillator or other implantable metallic device, epilepsy, stroke or recent head trauma);
* Patient who is not French-speaking or cannot read and write;
* Patient under guardianship;
* Patient in forced care (psychiatric care upon decision of the State representative and psychiatric care at the request of a third party);
* Pregnant woman or likely to be pregnant (of childbearing age) without effective contraception or breastfeeding;
* Patient participating in another clinical trial, or during a period of exclusion from another clinical trial;
* Patient who is not a beneficiary of a social security system.
* Patient who, according to the assessment of the investigator, risks not being compliant or diligent in the study procedures.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
average of the Scale for assessment of negative symptoms/scale for assessment of positive symptoms scale scores | 21 days
  The Primary Outcome Measure will be assessed by the average of the Scale for assessment of negative symptoms/scale for assessment of positive symptoms scale scores at approximately 21 days compared to the score at inclusion in the two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Rech, Montpellier, France